CLINICAL TRIAL: NCT07211893
Title: Effect of MyopiaEd Messaging on Improving Eye-use Behavior and Myopia Control Among Primary School Students in China: A Randomized Controlled Trial
Brief Title: Effect of MyopiaEd Messaging on Improving Eye-use Behavior and Myopia Control Among Primary School Students in China
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Collaborators: National Health Commission of the People's Republic of China (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025KYPJ113
Record Dates: First submitted 2025-09-18; First posted 2025-10-08 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MyopiaEd Messaging (Experimental): send myopia-related health education message from the MyopiaEd information repository
  Interventions: Other: Send myopia-related health education message
- Control (No Intervention): no myopia-related health education message from the MyopiaEd information repository

INTERVENTIONS:
Other: Send myopia-related health education message — Guardians of students in the intervention group will receive regular myopia-related health education messages, comprising text and images, from the MyopiaEd information repository via class-based WeChat groups. The intervention will last for 12 months.
  Arms: MyopiaEd Messaging

SUMMARY:
Myopia represents a significant global public health challenge, with China experiencing particularly high myopia prevalence among children and adolescents. The World Health Organization (WHO) acknowledges the critical role of health education in eye care and has collaborated with the International Telecommunication Union (ITU) to launch the Be He@lthy, Be Mobile (BHBM) initiative, which includes MyopiaEd-a mobile health project specifically designed to address myopia. Developed in partnership with international experts and informed by evidence-based guidelines, MyopiaEd provides standardized, scientifically validated content for effective myopia control. The MyopiaEd library has been translated and adapted by the Zhongshan Ophthalmic Center for use in China. Therefore, we aim to investigate whether the Chinese version of MyopiaEd can improve eye care behaviors among primary school students and enhance parental knowledge regarding myopia prevention and control in China.

ELIGIBILITY:
Inclusion Criteria:

* primary school students in the third grade;
* the guardians of students can receive, read, and understand multimedia (image-text) messages via WeChat on their mobile phones;
* voluntary participation in this study, with guardians' consent and a signed informed consent form.

Exclusion Criteria:

* with other ocular diseases that severely affect vision
* with systematic diseases or mental disorders, inability to understand or cooperate with the study

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1330 (Estimated)
Dates: Start 2025-12-05 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of children having improved eye-use behaviors after 1 year. | 12 months
  Children are considered to have improved behaviors if they meet three or more of the following criteria after 12 months:
  Outdoor Time: Increase of ≥ 30 minutes for those initially < 2 hours; maintain ≥ 2 hours for those initially ≥ 2 hours.
  Near Work Time: Reduce ≥ 30 minutes for those initially ≥ 1 hour; maintain < 1 hour for those initially < 1 hour.
  Screen Time: Reduce ≥ 30 minutes for those initially ≥ 1 hour; maintain < 1 hour for those initially < 1 hour.
  Eye Exam Frequency: Increase of ≥ 1 exam for those with < 2 exams initially; maintain ≥ 2 for those with ≥ 2 exams.
  Sitting Posture: Increase of ≥ 1 point for those with ≤ 3; maintain ≥ 4 for those with ≥ 4.
  Resting Behavior During Near Work: Increase of ≥ 1 point for those with ≤ 3; maintain ≥ 4 for those with ≥ 4.
  Spectacle-Wearing: Children not wearing glasses begin after 12 months. Daily Spectacle Wear for Myopic Children: Increase of ≥ 1 hour for those wearing ≤ 8 hours; maintain > 8 hours for those wearing > 8 hour.

SECONDARY OUTCOMES:
Change in myopia-related knowledge score of students' guardians between baseline and 12 months | 12 months
  Change in myopia-related knowledge score of students' guardians between baseline and 12 months, assessed via questionnaire. The score ranged from 1 to 20, with higher scores indicating better knowledge.
Difference in incidence of myopia between the two groups after 12 months | 12 months
  Difference in incidence of myopia between the two groups after 12 months
Difference in the change of spherical equivalence between baseline and 12 months in the two groups | 12 months
  Difference in the change of spherical equivalence between baseline and 12 months in the two groups. Spherical equivalence is calculated as sphere plus half of cylindrical power, as assessed by auto-refraction.
The satisfaction of the MyopiaEd information by the guardians | 12 months
  The satisfaction of the MyopiaEd information by the guardians, assessed by a study questionnaire. Satisfaction score ranges from 1 to 5, with higher scores indicating better satisfaction.

IPD SHARING:
Plan to Share IPD: No